CLINICAL TRIAL: NCT03052829
Title: Reducing Sedentary Time in Individuals With Pacemakers - Tracking By Pacemaker-Based Accelerometry
Brief Title: Physical Activity and Pacemaker Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Medtronic (Industry); University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Michael E. Widlansky, Associate Professor of Medicine and Pharmacology, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO27994
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Physical Activity; Pacemaker; Cardiovascular Diseases; Arrythmia
MeSH Terms: conditions — Motor Activity; Cardiovascular Diseases; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Activity Counseling (Experimental): Subjects will be given counseling on the benefits of increasing activity, instructions on how to slowly increase their activity over 12 weeks with walking, record their daily step counts, and have bi-weekly phone calls with study staff to reinforce the training and help them overcome barriers to being physically active.
  Interventions: Behavioral: Physical activity counseling
- Patient Usual Care (Placebo Comparator): Subjects will undergo usual care without intervention in this study arm
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Physical activity counseling — Subjects in this arm will receive counseling on how to increase their physical activity level.
  Arms: Physical Activity Counseling
Behavioral: Usual care — Subjects will undergo their usual care without intervention
  Arms: Patient Usual Care

SUMMARY:
The benefits of regular physical activity are well-established. Furthermore, the investigators have previously shown that in a population of patients with implanted pacemakers, those who exercise more than 2 hours daily have improved survival compared with those who exercise less than 2 hours daily. In this study, the aim f the investigators is to determine whether the offering subjects with pacemakers who have low levels of physical activity at baseline counseling to increase physical activity levels is effective as measured by their implanted device as well as by an external pacemaker.

The investigators seek to enroll about 30 patients into a 6-month 1:1 randomized interventional trial comparing the levels of physical activity in 2 groups, those who receive physical activity counseling versus usual care. The activity levels will be measured with external pedometers and with accelerometers embedded within the pacemaker device.

DETAILED DESCRIPTION:
The benefits of habitual physical activity (PA, activities of at least moderate intensity defined as ≥ 3 metabolic equivalents (METs)) are well-recognized. Emerging information from large data sets strongly suggest high levels of sedentary behavior, defined as activities <1.5 METs (equivalent to the amount of energy expended during seated activities such as computer work) increases the risk of diabetes, cardiovascular disease, and death, independent of the amount and intensity PA. The increased risk of sedentary behavior appears to be mediated at least in part by reduced insulin sensitivity, impaired lipid metabolism, increased vascular inflammation, and increased thrombotic tendencies.

The internal accelerometer embedded in Medtronic pacemakers registers, stores, and reports total number of "active time" based on a threshold activity intensity level of approximately 70 steps/min (estimated to be > 1.5 METs). This implanted accelerometer, combined with the regular follow-up required for appropriate care make individuals who have undergone Medtronic pacemaker implantation an ideal population in which to evaluate the impact of altering sedentary behavior on mortality and cardiovascular events.

The hypotheses are as follows:

1. a 12 week intervention to increase moderate intensity physical activity delivered at the point of care in patients with pacemakers will result in parallel increases in active time as measured by the pacemaker and step count as measured by pedometer.
2. the increase in activity measured by both the metrics in hypothesis 1 will be greater than with usual care.

Potential subjects who are interested in the study will have a screening visit to determine whether they meet the inclusion and exclusion criteria. Those who qualify and agree to participate will be randomized into either the Physical Activity Counseling arm (intervention arm) or the Patient Usual Care arm (control arm).

Subjects in the interventional arm will be given a pedometer and physical activity counseling on a regular basis for 3 months. Physical activity data from their external pedometer will be collected every 2 weeks via phone calls. Accelerometry data from the implanted pacemaker will be collected from the subject's medical record as pacemaker interrogations are performed every 3 months as part of routine clinical care. After the initial 3 month interventional phase is complete, these subjects will be followed for another 3 months with collection of pedometer as well as accelerometer data as described above.

Subjects in the control arm will be given pedometers for the week prior to pacemaker interrogation. These subjects will be called to report the number of steps they walked each day prior to the interrogation. Their accelerometry data will be captured through routine clinical pacemaker interrogations.

The primary outcome is the physical activity level in each group as measured by the accelerometer at time 0, 3 months and 6 months. The secondary outcome is the step count in each group as measured by the pedometer at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* Age > 55 years old
* Clinical indication for placement of permanent pacemaker
* LVEF of ≥ 50% at the time of or within 72 hours of implantation.
* Able to ambulate
* Average active time of ≤ 2 hours/day based on Revo or EnRhythm Accelerometery read out for the 3 month period prior to enrollment
* Able to take 650 steps over 10 minutes following pacemaker implantation (~2-2.5 mph walking speed)

Exclusion Criteria:

* Follow up for implantation planned at a non-study center at the time of implantation.
* Individuals with and expected life span of 1 year or less at the time of implantation
* Known history of cognitive impairment or inability to follow study procedures

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Widlansky, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin and Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Step-count data from the pedometers that the subjects wear along with the activity level as measured by the subject's pacemaker will be shared with the collaborating researchers at Medtronic and at UW-Milwaukee. This data will be obtained via phone conversations with the subject and via in-clinic or remote interrogations of the implanted pacemakers. The data will become available on an ongoing basis during the study duration as participants are contacted per the study protocol.

REFERENCES:
- [Derived] Puppala VK, Hofeld BC, Anger A, Tyagi S, Strath SJ, Fox J, Berger MG, Ahn KW, Widlansky ME. Pacemaker detected active minutes are superior to pedometer-based step counts in measuring the response to physical activity counseling in sedentary older adults. BMC Geriatr. 2020 May 6;20(1):162. doi: 10.1186/s12877-020-01559-y. PMID 32375676

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physical Activity Counseling | Patient Usual Care
Started | 11 | 10
Completed | 7 | 6
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Activity Counseling | Patient Usual Care | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 84 (5) | 75 (5) | 80 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 30.0 (5.0) | 32.5 (6.6) | 31.2 (5.7)
History of Sustained Ventricular Tachycardia [Count of Participants; unit: Participants] | 0 | 3 | 3
History of Non-Sustained Ventricular Tachycardia [Count of Participants; unit: Participants] | 2 | 5 | 7
Sick Sinus Syndrome [Count of Participants; unit: Participants] | 1 | 3 | 4
High Degree AV Block [Count of Participants; unit: Participants] | 6 | 3 | 9
Creatinine Clearance < 60 mL/min/1.73 m2 [Count of Participants; unit: Participants] | 4 | 1 | 5
Hypertension [Count of Participants; unit: Participants] | 6 | 4 | 10
Hyperlipidemia [Count of Participants; unit: Participants] | 6 | 6 | 12
Diabetes [Count of Participants; unit: Participants] | 0 | 3 | 3
Heart Failure [Count of Participants; unit: Participants] | 0 | 2 | 2
Coronary Stent [Count of Participants; unit: Participants] | 1 | 0 | 1
Prior CABG [Count of Participants; unit: Participants] | 1 | 0 | 1
Prior CVA [Count of Participants; unit: Participants] | 1 | 4 | 5
Atrial Fibrillation [Count of Participants; unit: Participants] | 3 | 4 | 7
LVEF% [Mean (Standard Deviation); unit: %] | 62 (3) | 57 (4) | 60 (4)
LV End Diastolic Dimension [Mean (Standard Deviation); unit: mm] | 43 (3) | 44 (6) | 44 (5)
LV End Systolic Dimension [Mean (Standard Deviation); unit: mm] | 26 (2) | 30 (9) | 28 (6)
Percent Atrial Pacing [Mean (Standard Deviation); unit: %] | 66 (31) | 53 (38) | 61 (34)
Percent Ventricular Pacing [Mean (Standard Deviation); unit: %] | 12 (21) | 34 (51) | 22 (38)
Moderate or Greater Mitral Regurgitation [Count of Participants; unit: Participants] | 2 | 0 | 2
Current Smoker [Count of Participants; unit: Participants] | 0 | 1 | 1
ACEI or ARB Therapy [Count of Participants; unit: Participants] | 3 | 4 | 7
Beta Blocker Therapy [Count of Participants; unit: Participants] | 4 | 3 | 7
HMG CoA Reductase Therapy [Count of Participants; unit: Participants] | 4 | 4 | 8
SBP [Mean (Standard Deviation); unit: mmHg] | 131 (27) | 121 (14) | 126 (22)
DBP [Mean (Standard Deviation); unit: mmHg] | 70 (9) | 77 (18) | 73 (14)
HR [Mean (Standard Deviation); unit: bpm] | 66 (4) | 70 (7) | 68 (6)
Calculated Gait Speed [Mean (Standard Deviation); unit: m/sec] | 0.84 (0.14) | 0.86 (0.18) | 0.85 (0.16)
Pacemaker detected active minutes [Mean (Standard Deviation); unit: hours/day] | 1.59 (0.44) | 1.62 (0.18) | 1.60 (0.33)
Pedometer-Based Daily Step Count [Mean (Standard Deviation); unit: steps/day] | 2827 (1641) | 2474 (1623) | 2618 (1594)

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity Level as Measured by Embedded Accelerometer
Description: This is the daily measured active hours in the device
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: active hours/day
Arm/Group | Physical Activity Counseling | Patient Usual Care
Number analyzed (Participants) | 7 | 6
active hours/day | 1.97 (0.56) | 1.77 (0.22)

2. Secondary Outcome: Physical Activity Level as Measured by External Pedometer
Description: this is a daily step count (one week average)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Physical Activity Counseling | Patient Usual Care
Number analyzed (Participants) | 7 | 6
steps/day | 1769 (771) | 2487 (1800)

ADVERSE EVENTS:
Time Frame: Information on adverse events were recorded over the 1st 12 weeks of the study which contained the intervention
Arm/Group | Physical Activity Counseling | Patient Usual Care
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
Unable to complete projected enrollment due to difficulties with recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT03052829/Prot_SAP_000.pdf